CLINICAL TRIAL: NCT04640740
Title: Isokinetic Performance and Function Are Similar 12 Months After Total Hip Arthroplasty Applied With a Posterior or Anterolateral Approach: A Randomized Controlled Trial
Brief Title: Isokinetic Performance and Function After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Deniz CANKAYA, Assoc. Professor, Gulhane Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-17-1415
Record Dates: First submitted 2020-11-18; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Hip Osteoarthritis
Keywords: anterolateral approach; posterior approach; isokinetic test
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anterolateral approach (ALA) (Experimental): anterolateral surgical approach of total hip arthroplasty
  Interventions: Procedure: hip arthroplasty
- posterior approach (PA) (Experimental): posterior surgical approach of total hip arthroplasty.
  Interventions: Procedure: hip arthroplasty

INTERVENTIONS:
Procedure: hip arthroplasty — two different approaches of total hip arthroplasty

SUMMARY:
There are ongoing debates on the effects of the surgical approach on outcome after total hip arthroplasty. It was hypothesized that with the anterolateral approach, trauma to the abductor arm can be occured and related detrimental effects can diminish the post-operative outcomes. In this first randomized controlled trial in the literature on this subject, isokinetic performance and patient-reported functional outcomes were evaluated in patients undergoing total hip arthroplasty. with a posterior approach (PA) and a anterolateral approach (ALA), at 6 and 12 months postoperatively.

DETAILED DESCRIPTION:
Patients undergoing total hip arthroplasty are randomized to posterior approach (PA) and anterolateral approach (ALA) groups. The patients are evaluated preoperatively and at 6 and 12 months postoperatively, with flexion, extension and abduction strength measurements and the Harris Hip Score (HHS). The physiatrist performing isokinetic tests and the patients are blinded to the study groups.All data are calculated as mean and standard deviation values. The Student's t-test is used for statistical analysis of the patient data. Statistical calculations are performed using SPSS vn.22.0 software (IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

Patients aged 55 to 80 years unilateral primary hip osteoarthritis -

Exclusion Criteria:

bilateral osteoarthritis inflammatory arthritis post-traumatic osteoarthritis previous hip surgery neuromuscular diseases

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
isokinetic test | Change from preoperative isokinetic test results at 6th months and 12th months isokinetic test results
  isokinetic test during flexion, extension and abduction of the hip

SECONDARY OUTCOMES:
Harris Hip Score | Change from preoperativeHarris Hip Score results at 6th months and 12th months iHarris Hip Score results
  Functional score of the hip. Harris Hip Score: 100-90: Excellent 89-80:Good 79-70:Fair below 70:Poor

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane Teaching and Research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Cankaya D, Inci F, Karakus D, Turker HB, Kahve Y, Neyisci C. Isokinetic performance and function are similar after total hip arthroplasty applied with a posterior or anterolateral approach: a randomised controlled trial. Hip Int. 2023 Jan;33(1):67-72. doi: 10.1177/11207000211012989. Epub 2021 Apr 26. PMID 33896243